CLINICAL TRIAL: NCT04347629
Title: Improving Medical Decision Making for Older Patients With End Stage Renal Disease
Acronym: VIDEO-KD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-39981; 1R01AG066892 (NIH)
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Renal Disease, End Stage; Palliative Care; Decision Aids
Keywords: video decision aid; video declaration; aging population
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Usual clinical care
- Video Decision Aid (Experimental): The video intervention consists of a video decision aid along with a video declaration (ViDec), which is recorded by the patient. The video decision aid explores ACP options for medical care for end-stage renal disease (ESRD) and reviews hemodialysis, peritoneal dialysis, as well as medical management without dialysis; it also reviews cardiopulmonary resuscitation (CPR). Patients will also audio- or video-record their preferences using a tablet.
  Interventions: Behavioral: Advance Care Planning Video Decision Aid

INTERVENTIONS:
Behavioral: Advance Care Planning Video Decision Aid — The video decision aid explores ACP options for medical care for end-stage renal disease (ESRD) and reviews hemodialysis, peritoneal dialysis, as well as medical management without dialysis; it also reviews cardiopulmonary resuscitation (CPR). Patients will also audio- or video-record their preferences using a tablet.
  Arms: Video Decision Aid

SUMMARY:
The overall objective of this study is to reduce the burden of chronic kidney disease (CKD) and its consequences for an aging U.S. population. To accomplish this, the investigators propose to conduct a multi-center randomized trial of an advance care planning (ACP) video intervention (vs. usual care) among older patients with CKD.

DETAILED DESCRIPTION:
The video intervention consists of a video decision aid along with a video declaration (ViDec), which is recorded by the patient. The video decision aid explores ACP options for medical care for end-stage renal disease (ESRD) and reviews hemodialysis, peritoneal dialysis, as well as medical management without dialysis; it also reviews cardiopulmonary resuscitation (CPR). Patients will also audio- or video-record their preferences using a tablet. The video will be shared with their nephrologist. The patient will have a copy of the video to take with them and share with their loved ones.

Patients will answer survey questions about their preferences, knowledge, decisional conflict, and ACP engagement. They will be surveyed every two months for one year or death (if they die before one year).

Potential participants will be recruited from 10 nephrology clinics: Massachusetts General Hospital (n=75), Brigham and Women's Hospital (n=75), University of Pittsburgh (n=75), University of Pennsylvania, Stanford University, Palo Alto Veterans Institute for Research, University of Washington, Renal & Transplant Associates of New England, University of New Mexico and Boston Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥70 are eligible if they have EITHER Advanced CKD defined as ONE eGFR value ≤ 30 ml/min/1.73m2 in the past 12 months NOT determined to be a result of AKI OR Have a diagnosis of CKD and less than a two-year prognosis from any cause, defined by the clinician answering "NO" to the Surprise Question ("Would you be surprised if this patients died in the next two years?")
* Patients age 65-69 are eligible if they have BOTH Advanced CKD defined as ONE eGFR value ≤ 30 ml/min/1.73m2 NOT determined to be a result of AKI AND Have less than a two-year prognosis, defined by the clinician answering "NO" to the Surprise Question ("Would you be surprised if this patients died in the next two years?")
* Patients who have not had a nephrology visit in the past 12 months can be recruited from non-Nephrology Clinics per the above eligibility criteria

Exclusion Criteria:

* listed for kidney transplantation or previous transplant recipient
* already on or previously on dialysis (including emergent dialysis)
* new patient visit
* visually impaired beyond 20/200 corrected
* psychological state not appropriate for ACP discussions as determined by the primary nephrologist
* cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 456 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Advance Care Planning (ACP) in Electronic Health Record (EHR) Documentation | Baseline, 12 months
  Documentation in the electronic health record reflecting an ACP conversation (any of the following: completion of advance directive or physician order for life sustaining treatment (POLST); code status documentation; provider note reflecting ACP discussion).

SECONDARY OUTCOMES:
Change in ACP Engagement | baseline, 12 months
  4 investigator designed questions about actions patient has taken with regards to ACP
Change in ACP Preferences | Baseline, 12 months
  survey assessment
Change in ACP Conversations | Baseline, 12 months
  3 investigator designed questions about conversations with family/friends about ACP
Change in Kidney Disease (KD) Specific Quality of Life (QOL) | Baseline, 12 months
  KD-QOL is a validated instrument to assess QOL that includes 36 questions with response options in likert scale format. The outcome measure is the difference in averaged scores between baseline and 12 months; It is calculated as (Score at visit 2 - Score at visit 1).
  QOL is assessed by three components; physical health score, mental health score and kidney disease health score. Physical health score, mental health score and kidney disease health score are averaged scores of sub-scales. The range of each score and each sub-scale are 0 - 100, and higher values indicate better QOL status.
Change in Health Related Quality of Life (QoL) | Baseline, 12 months
  Health related quality of life will be assessed using a validated instrument EuroQol-5D (EQ-5D) which has two components. There is a descriptive system with 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. the other component is a visual analogue scale (VAS) that records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
Change in Decisional Conflict | Baseline, 12 months
  We will measure decisional conflict using the decisional conflict scale (DCS), which attempts to measure decisional uncertainty.
Acceptability of video intervention | Baseline
  For those patients randomized to the video intervention, we will measure, via survey, acceptability of the decision aid using a modified version of the validated Yorkshire Dialysis Decision Aid Usefulness Scale. We will also ask questions regarding comfort viewing the video, which we have validated in our prior work.
Change in CKD Care Preferences | Baseline, 12 months
  All patients will be asked their preferences for kidney failure care at baseline. We will then assess their follow-up preferences by chart review in the electronic medical record.
Healthcare Costs | Baseline, 12 months
  We will identify the major components of healthcare services used, including inpatient, pharmacy, outpatient, emergency department and dialysis. We will also examine utilization by subgroups with comorbidity of diabetes, heart failure and cardiovascular disease. We will use Medicare claims data to obtain the associated costs, including payments by Medicare and secondary payers (e.g., out-of-pocket payments).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Paasche-Orlow, MD, MPH, Principal Investigator — Tufts Medical Center
Locations (9):
- United States (9):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University, Palo Alto, California
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
  - The University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The phenotypic data associated with enrolled participants will be shared by depositing these data in the Open Science Framework data repository. Additional data documentation and de-identified IPD including demographics, diagnoses, and outcomes will be deposited. Resources such as study protocols and statistical analysis codes will also be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Outcome data will be deposited into Open Science Framework repository as soon as possible but no later than within one year of the completion of the funded project period for the parent award or upon acceptance of the data for publication, or public disclosure of a submitted patent application, whichever is earlier. Data will remain available for a period of 5 years.
Access Criteria: Data and supporting information will be shared with investigators working in accordance to guidelines set by the data repository. Meta-analysis data and associated phenotypic data, along with data content, format, and organization, will be made available to investigators through the Open Science Framework data repository.

REFERENCES:
- [Derived] Eneanya ND, Lakin JR, Paasche-Orlow MK, Lindvall C, Moseley ET, Henault L, Hanchate AD, Mandel EI, Wong SPY, Zupanc SN, Davis AD, El-Jawahri A, Quintiliani LM, Chang Y, Waikar SS, Bansal AD, Schell JO, Lundquist AL, Tamura MK, Yu MK, Unruh ML, Argyropoulos C, Germain MJ, Volandes A. Video Images about Decisions for Ethical Outcomes in Kidney Disease (VIDEO-KD): the study protocol for a multi-centre randomised controlled trial. BMJ Open. 2022 Apr 8;12(4):e059313. doi: 10.1136/bmjopen-2021-059313. PMID 35396311